CLINICAL TRIAL: NCT04540432
Title: Descriptive Study on the Evolution of Intestinal Microbiota Profiles in Patients With Juvenile Spondylarthropathy According to the Typology of Treatment and Response to it: A Descriptive, Prospective Pilot Study
Brief Title: Evolution of Intestinal Microbiota in Patients With Juvenile Spondylarthropathy According to Typology of Treatment
Acronym: MESAJ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University Hospital, Montpellier (Other); Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIMAO/2019/TAT-01; 20.03.20.564 (Other: CNRIPH)
Record Dates: First submitted 2020-08-27; First posted 2020-09-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Spondylarthropathies
Keywords: Microbiota
MeSH Terms: conditions — Spondylarthropathies | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Patients will be split into 4 groups according to their treatment profile:
  Profile A = patients on non-steroidal anti-inflammatory drugs.
  Profile AM = patients on non-steroidal anti-inflammatory drugs followed by treatment with methotrexate until the end of the study.
  Profile AB = patients on non-steroidal anti-inflammatory drugs, followed by biotherapy until the end of the study.
  Profile AMB = patients on non-steroidal anti-inflammatory drugs followed by treatment with methotrexate and then biotherapy until the end of the study.
  Profile M : methotrexate alone
  Profile B : biothérapy alone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Profile AB (Experimental): Patients on non-steroidal anti-inflammatory drugs followed by biotherapy.
  Interventions: Other: Stool collection at the patient's home.; Diagnostic Test: Blood test
- Profile AM (Experimental): Patients on non-steroidal anti-inflammatory drugs followed by treatment with methotrexate.
  Interventions: Other: Stool collection at the patient's home.; Diagnostic Test: Blood test
- Profile AMB (Experimental): Patients on non-steroidal anti-inflammatory drugs followed by treatment with methotrexate and then biotherapy if there is no improvement with methotrexate.
  Interventions: Other: Stool collection at the patient's home.; Diagnostic Test: Blood test
- Profile A (Experimental): Patients on non-steroidal anti-inflammatory drugs.
  Interventions: Other: Stool collection at the patient's home.; Diagnostic Test: Blood test
- Profile M (Experimental): methotrexate alone
  Interventions: Other: Stool collection at the patient's home.; Diagnostic Test: Blood test
- Profile B (Experimental): biotherapy alone
  Interventions: Other: Stool collection at the patient's home.; Diagnostic Test: Blood test

INTERVENTIONS:
Other: Stool collection at the patient's home. — Stool samples will be taken from each patient to look for changes in intestinal microbiota. These collections will be made on Day 0 +24h, 24 hours before the 1st follow-up visit after 1 month of treatment with non-steroidal anti-inflammatory drugs, 24 hours after the second follow-up visit (between months 3 and 4) and finally, at the end of treatment.
Diagnostic Test: Blood test — 7 ml of blood will be taken from each patient before treatment i.e. at the inclusion visit and at the end of treatment.

SUMMARY:
Idiopathic juvenile arthritis includes 20% of patients with arthritis with enthesitis or juvenile spondyloarthropathy. This is treated with anti-inflammatory drugs and then followed by biotherapy with DMARDs (Drugs Modifying the Activity of Rheumatic Disease) if the former are insufficient. Methotrexate (MTX) may also be used before these biotherapies. Recently, in adults, a particular profile of intestinal microbiota has been shown to alter the availability of MTX making it in efficient. Knowing that pediatric patients with juvenile spondyloarthropathy have an imbalance of their intestinal flora (dysbiosis) the investigators wanted to explore whether DMARDs could have a similar impact on the microbiota of these young patients and alter the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 6 and under 17 years old (included).
* Patients diagnosed with arthritis with juvenile enthesitis according to the International League of Associations for Rheumatology (ILAR) criteria.
* Patients who haven't been treated by Methotrexate or biotherapy for at least 3 months.
* Patients who haven't been treated by cortisone for over a month.
* Patients whose parents have given written informed consent.
* Patients for whom the consent form has been signed by their legal guardian.
* Patients covered by the Social Security System or benefitting from private health insurance.

Exclusion Criteria:

* Patients enrolled in another category 1 study or who have already taken part in a category 1 study within 3 months prior to inclusion.
* Patients who are within an exclusion period determined by another study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2029-06-28 (Estimated); Study Completion 2029-06-28 (Estimated)

PRIMARY OUTCOMES:
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A). Number of species detected in the intestinal microbiota. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A). Distribution of species detected in the intestinal microbiota. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The distribution of the various bacterial species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A). Diversity of species detected in the intestinal microbiota. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The diversity index according to the number of species and the number of functional groups will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A). Number of species detected in the intestinal microbiota. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The number of species detected in the intestinal microbiota will be recorded.
  - the diversity index according to the number of species and the number of functional groups.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A). Distribution of species detected in the intestinal microbiota. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The distribution of the various bacterial species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A). Diversity of species detected in the intestinal microbiota. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The diversity index according to the number of species and the number of functional groups will be recorded.
Response to treatment in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A) | After 1 month of treatment
  The JADAS CRP clinical score will be used to rate the degree of activity of the disease. The Juvenile Arthritis Disease Activity Score (JADAS) is a recently developed composite tool for scoring disease activity in juvenile idiopathic arthritis. It is a composite disease activity score including four measures:
  * the physician's global assessment of disease activity;
  * the parent/guardian's or patient's global assessment of overall wellbeing;
  * number of joints with active arthritis; and
  * C-reactive protein (CRP) which has been determined as an alternative inflammatory marker to the Erythrocyte Sedimentation Rate ESR. JADAS-CRP was calculated similarly to the original JADAS as the simple sum of its four components, yielding a global score of 0-40, 0-57 and 0-101 depending on the joint count used for the JADAS10-CRP, JADAS27-CRP and JADAS71-CRP, respectively.
Response to treatment in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A). Number of flare-ups. | After 1 month of treatment
  The number of flare-ups in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A) will be noted.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM). Number of species detected in the intestinal microbiota. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM). Distribution of species detected in the intestinal microbiota. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The distribution of the various bacterial species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM). Diversity of species detected in the intestinal microbiota. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The diversity index according to the number of species and the number of functional groups will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM).Number of species. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM). Distribution of species. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The distribution of the various bacterial species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM). Diversity of species. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The diversity index according to the number of species and the number of functional groups will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM). Number of species. | After 6 months of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM). Distribution of species. | After 6 months of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The distribution of the various bacterial species in the microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM). Diversity of species. | After 6 months of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The diversity index according to the number of species and the number of functional groups will be recorded.
Response to treatment in patients treated with non-steroidal anti-inflammatory drugs for 1 month followed by methotrexate for 5 months (Profile AM) | After 6 months of treatment
  The JADAS CRP clinical score will be used to rate the degree of activity of the disease. The Juvenile Arthritis Disease Activity Score (JADAS) is a recently developed composite tool for scoring disease activity in juvenile idiopathic arthritis. It is a composite disease activity score including four measures:
  * the physician's global assessment of disease activity;
  * the parent/guardian's or patient's global assessment of overall wellbeing;
  * number of joints with active arthritis; and
  * C-reactive protein (CRP) which has been determined as an alternative inflammatory marker to the Erythrocyte Sedimentation Rate ESR. JADAS-CRP was calculated similarly to the original JADAS as the simple sum of its four components, yielding a global score of 0-40, 0-57 and 0-101 depending on the joint count used for the JADAS10-CRP, JADAS27-CRP and JADAS71-CRP, respectively.
Response to treatment in patients treated with non-steroidal anti-inflammatory drugs for 1 month followed by methotrexate for 5 months (Profile AM). Number of flare-ups. | After 6 months of treatment
  The number of flare-ups in patients treated with non-steroidal anti-inflammatory drugs for 1 month followed by methotrexate for 5 months (Profile AM) will be noted.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Number of species. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Distribution of species. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The distribution of the various bacterial species in the microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Diversity of species. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The diversity index according to the number of species and the number of functional groups will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Number of species. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Distribution of species. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The distribution of the various bacterial species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Diversity of species. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The diversity index according to the number of species and the number of functional groups will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Number of species. | After 6 months of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Distribution of species. | After 6 months of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The distribution of the various bacterial species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Diversity of species. | After 6 months of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The diversity index according to the number of species and the number of functional groups will be recorded.
Response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB) | After 6 months of treatment
  The JADAS CRP clinical score will be used to rate the degree of activity of the disease. The Juvenile Arthritis Disease Activity Score (JADAS) is a recently developed composite tool for scoring disease activity in juvenile idiopathic arthritis. It is a composite disease activity score including four measures:
  * the physician's global assessment of disease activity;
  * the parent/guardian's or patient's global assessment of overall wellbeing;
  * number of joints with active arthritis; and
  * C-reactive protein (CRP) which has been determined as an alternative inflammatory marker to the Erythrocyte Sedimentation Rate ESR. JADAS-CRP was calculated similarly to the original JADAS as the simple sum of its four components, yielding a global score of 0-40, 0-57 and 0-101 depending on the joint count used for the JADAS10-CRP, JADAS27-CRP and JADAS71-CRP, respectively.
Response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB). Number of flare-ups. | After 6 months of treatment
  The number of flare-ups in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB) will be noted.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Number of species. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Distribution of species. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The distribution of the various bacterial species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Diversity of species. | 24 hours after inclusion
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department.The diversity index according to the number of species and the number of functional groups will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Number of species. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Distribution of species. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The distribution of the various bacterial species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Diversity of species. | After 1 month of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The diversity index according to the number of species and the number of functional groups will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Number of species. | After 6 months of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The number of species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Distribution of species. | After 6 months of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The distribution of the various bacterial species detected in the intestinal microbiota will be recorded.
Evolution of the intestinal microbiota in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Diversity of species. | After 6 months of treatment
  Patients will provide 2 stool samples (one for analysis and one for the biobank) taken at the patient's home, preserved at -20°C and transported in a coolerbag to the hospital. One sample will be frozen to -80°C for the biobank and one sample will be kept at -20°C at the pediatric department. The diversity index according to the number of species and the number of functional groups will be recorded.
Response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB) | After 6 months of treatment
  The JADAS CRP clinical score will be used to rate the degree of activity of the disease. The Juvenile Arthritis Disease Activity Score (JADAS) is a recently developed composite tool for scoring disease activity in juvenile idiopathic arthritis. It is a composite disease activity score including four measures:
  * the physician's global assessment of disease activity;
  * the parent/guardian's or patient's global assessment of overall wellbeing;
  * number of joints with active arthritis; and
  * C-reactive protein (CRP) which has been determined as an alternative inflammatory marker to the Erythrocyte Sedimentation Rate ESR. JADAS-CRP was calculated similarly to the original JADAS as the simple sum of its four components, yielding a global score of 0-40, 0-57 and 0-101 depending on the joint count used for the JADAS10-CRP, JADAS27-CRP and JADAS71-CRP, respectively.
Response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB). Number of flare-ups. | After 6 months of treatment
  The number of flare-ups in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB) will be noted.

SECONDARY OUTCOMES:
A:Correlation between intestinal microbiota of patients treated with non-steroidal anti-inflammatory drugs alone (Profile A) and the clinical stage of evolution of Juvenile Spondylarthitis. | 24 hours after inclusion
  The description of the intestinal microbiota profile according to INSERM laboratory Unit 1047 will be correlated with the clinical stage of the disease (on remission or acute flare) before and after treatment.
A:Correlation between intestinal microbiota of patients treated with non-steroidal anti-inflammatory drugs alone (Profile A) and the clinical stage of evolution of Juvenile Spondylarthitis. | After 1 month of treatment
  The description of the intestinal microbiota profile according to INSERM laboratory Unit 1047 will be correlated with the clinical stage of the disease (on remission or acute flare) before and after treatment.
A:Correlation between intestinal microbiota of patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM) and the clinical stage of evolution of Juvenile Spondylarthitis. | 24 hours after inclusion
  The description of the intestinal microbiota profile according to INSERM laboratory Unit 1047 will be correlated with the clinical stage of the disease (on remission or acute flare) before and after treatment.
A:Correlation between intestinal microbiota of patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM) and the clinical stage of evolution of Juvenile Spondylarthitis. | After 6 months of treatment
  The description of the intestinal microbiota profile according to INSERM laboratory Unit 1047 will be correlated with the clinical stage of the disease (on remission or acute flare) before and after treatment.
A:Correlation between intestinal microbiota of patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB) and the clinical stage of evolution of Juvenile Spondylarthitis. | 24 hours after inclusion
  The description of the intestinal microbiota profile according to INSERM laboratory Unit 1047 will be correlated with the clinical stage of the disease (on remission or acute flare) before and after treatment.
A: Correlation between intestinal microbiota of patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB) and the clinical stage of evolution of Juvenile Spondylarthitis. | After 6 months of treatment
  The description of the intestinal microbiota profile according to INSERM laboratory Unit 1047 will be correlated with the clinical stage of the disease (on remission or acute flare) before and after treatment.
A:Correlation between intestinal microbiota of patients treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy (Profile AMB) and the clinical stage of evolution of Juvenile Spondylarthitis. | 24 hours after inclusion
  The description of the intestinal microbiota profile according to INSERM laboratory Unit 1047 will be correlated with the clinical stage of the disease (on remission or acute flare) before and after treatment.
A:Correlation between intestinal microbiota of patients treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy (Profile AMB) and the clinical stage of evolution of Juvenile Spondylarthitis. | After 6 months of treatment
  The description of the intestinal microbiota profile according to INSERM laboratory Unit 1047 will be correlated with the clinical stage of the disease (on remission or acute flare) before and after treatment.
B:Correlation between bacterial translocation and response to treatment in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A) | 24 hours after inclusion
  Pre- and post-therapeutic translocation and response to treatment (presence/absence: detection of DNA 16S in the blood, quantification by quantitative PCR and sequencing for identification).
B:Correlation between bacterial translocation and response to treatment in patients treated with non-steroidal anti-inflammatory drugs alone (Profile A) | After 1 month of treatment
  Pre- and post-therapeutic translocation and response to treatment (presence/absence: detection of DNA 16S in the blood, quantification by quantitative PCR and sequencing for identification).
B:Correlation between bacterial translocation and response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM) | 24 hours after inclusion
  Pre- and post-therapeutic translocation and response to treatment (presence/absence: detection of DNA 16S in the blood, quantification by quantitative PCR and sequencing for identification).
B:Correlation between bacterial translocation and response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate (Profile AM) | After 6 months of treatment
  Pre- and post-therapeutic translocation and response to treatment (presence/absence: detection of DNA 16S in the blood, quantification by quantitative PCR and sequencing for identification).
B:Correlation between bacterial translocation and response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB) | 24 hours after inclusion
  Pre- and post-therapeutic translocation and response to treatment (presence/absence: detection of DNA 16S in the blood, quantification by quantitative PCR and sequencing for identification).
B:Correlation between bacterial translocation and response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by biotherapy (Profile AB) | After 6 months of treatment
  Pre- and post-therapeutic translocation and response to treatment (presence/absence: detection of DNA 16S in the blood, quantification by quantitative PCR and sequencing for identification).
B:Correlation between bacterial translocation and response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB) | 24 hours after inclusion
  Pre- and post-therapeutic translocation and response to treatment (presence/absence: detection of DNA 16S in the blood, quantification by quantitative PCR and sequencing for identification).
B:Correlation between bacterial translocation and response to treatment in patients treated with non-steroidal anti-inflammatory drugs followed by methotrexate then biotherapy (Profile AMB) | After 6 months of treatment
  Pre- and post-therapeutic translocation and response to treatment (presence/absence: detection of DNA 16S in the blood, quantification by quantitative PCR and sequencing for identification).
C:Constitution of a biobank of samples from Profile A patients (treated with non-steroidal anti-inflammatory drugs alone) | After 6 months of treatment
  All blood and stool samples used for the study will be deposited in the biobank for reference.
C: Constitution of a biobank for Profile AM patients (treated with non-steroidal anti-inflammatory drugs then methotrexate). | After 6 months of treatment
  All blood and stool samples used for the study will be deposited in the biobank for reference.
C: Constitution of a biobank for Profile AB patients (treated with non-steroidal anti-inflammatory drugs then biotherapy) | At the inclusion visit on Day 0
  All blood and stool samples used for the study will be deposited in the biobank for reference.
C: Constitution of a biobank for AMB patients (treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy) | At the inclusion visit on Day 0
  All blood and stool samples used for the study will be deposited in the biobank for reference.
Age of Profile A patients (treated with non-steroidal anti-inflammatory drugs alone) | At the inclusion visit on Day 0
  Recorded in years
Weight of Profile A patients (treated with non-steroidal anti-inflammatory drugs alone) | At the inclusion visit on Day 0
  Recorded in kilos
Height of Profile A patients (treated with non-steroidal anti-inflammatory drugs alone) | At the inclusion visit on Day 0
  Recorded in cm.
Sex of Profile A patients (treated with non-steroidal anti-inflammatory drugs alone) | At the inclusion visit on Day 0
  Male/Female
Previous treatment in Profile A patients (treated with non-steroidal anti-inflammatory drugs alone) | At the inclusion visit on Day 0
  The investigators will record details of all treatment followed prior to diagnosis of juvenile spondylarthritis:
  * NSAIDs : dosage and dates
  * Corticoids : dosage and dates
  * Antibiotics : dosage and dates
  * DMARDs : dosage and dates
Dietary habits in Profile A patients (treated with non-steroidal anti-inflammatory drugs alone) | At the inclusion visit on Day 0
  The investigators will record details of patients' dietary habits and, more particularly, note all foods which are excluded.
Food allergies in Profile A patients (treated with non-steroidal anti-inflammatory drugs alone) | At the inclusion visit on Day 0
  The investigators will record details of patients' food allergies.
Lifestyle of Profile A patients (treated with non-steroidal anti-inflammatory drugs alone) | At the inclusion visit on Day 0
  The investigators will record details of the patient's lifestyle:
  * Brothers and sisters (number and date of birth of each one)
  * Communities (date of entry)
  * Contact with animals
Age of Profile AM patients (treated with non-steroidal anti-inflammatory drugs then methotrexate) | At the inclusion visit on Day 0
  Recorded in years
Weight of Profile AM patients (treated with non-steroidal anti-inflammatory drugs then methotrexate) | At the inclusion visit on Day 0
  Recorded in kilos
Height of Profile AM patients (treated with non-steroidal anti-inflammatory drugs then methotrexate) | At the inclusion visit on Day 0
  Recorded in cm.
Sex of Profile AM patients (treated with non-steroidal anti-inflammatory drugs then methotrexate) | At the inclusion visit on Day 0
  Male/Female
Previous treatment in Profile AM patients (treated with non-steroidal anti-inflammatory drugs then methotrexate) | At the inclusion visit on Day 0
  The investigators will record details of all treatment followed prior to diagnosis of juvenile spondylarthritis:
  * NSAIDs : dosage and dates
  * Corticoids : dosage and dates
  * Antibiotics : dosage and dates
  * DMARDs : dosage and dates
Dietary habits in Profile AM patients (treated with non-steroidal anti-inflammatory drugs then methotrexate) | At the inclusion visit on Day 0
  The investigators will record details of all patients' dietary habits and, more particularly, note all foods which are excluded.
Food allergies in Profile AM patients (treated with non-steroidal anti-inflammatory drugs then methotrexate) | At the inclusion visit on Day 0
  The investigators will record details of all patients' food allergies.
Lifestyle in Profile AM patients (treated with non-steroidal anti-inflammatory drugs then methotrexate) | At the inclusion visit on Day 0
  The investigators will record details of the patient's lifestyle:
  * Brothers and sisters (number and date of birth of each one)
  * Communities (date of entry)
  * Contact with animals
Age of Profile AB patients (treated with non-steroidal anti-inflammatory drugs then biotherapy) | At the inclusion visit on Day 0
  Recorded in years
Weight of Profile AB patients (treated with non-steroidal anti-inflammatory drugs then biotherapy) | At the inclusion visit on Day 0
  Recorded in kilos
Height of Profile AB patients (treated with non-steroidal anti-inflammatory drugs for then biotherapy) | At the inclusion visit on Day 0
  Recorded in cm.
Sex of Profile AB patients (treated with non-steroidal anti-inflammatory drugs then biotherapy) | At the inclusion visit on Day 0
  Male/Female
Previous treatment in Profile AB patients (treated with non-steroidal anti-inflammatory drugs then biotherapy) | At the inclusion visit on Day 0
  The investigators will record details of all treatment followed prior to diagnosis of juvenile spondylarthritis:
  * NSAIDs : dosage and dates
  * Corticoids : dosage and dates
  * Antibiotics : dosage and dates
  * DMARDs : dosage and dates
Dietary habits in Profile AB patients (treated with non-steroidal anti-inflammatory drugs then biotherapy) | At the inclusion visit on Day 0
  The investigators will record details of all patients' dietary habits and, more particularly, note all foods which are excluded.
Food allergies in Profile AB patients (treated with non-steroidal anti-inflammatory drugs then biotherapy) | At the inclusion visit on Day 0
  The investigators will record details of all patients' food allergies.
Lifestyle in Profile AB patients (treated with non-steroidal anti-inflammatory drugs then biotherapy) | At the inclusion visit on Day 0
  The investigators will record details of the patient's lifestyle:
  * Brothers and sisters (number and date of birth of each one)
  * Communities (date of entry)
  * Contact with animals
Age of Profile AMB patients (treated with non-steroidal anti-inflammatory drugs then methotrexate biotherapy) | At the inclusion visit on Day 0
  Recorded in years
Weight of Profile AMB patients (treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy) | At the inclusion visit on Day 0
  Recorded in kilos
Height of Profile AMB patients (treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy) | At the inclusion visit on Day 0
  Recorded in cm.
Sex of Profile AMB patients (treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy) | At the inclusion visit on Day 0
  Male/Female
Previous treatment in Profile AMB patients (treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy) | At the inclusion visit on Day 0
  The investigators will record details of all treatment followed prior to diagnosis of juvenile spondylarthritis:
  * NSAIDs : dosage and dates
  * Corticoids : dosage and dates
  * Antibiotics : dosage and dates
  * DMARDs : dosage and dates
Dietary habits in Profile AMB patients (treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy) | At the inclusion visit on Day 0
  The investigators will record details of all patients' dietary habits and, more particularly, note all foods which are excluded.
Food allergies in Profile AMB patients (treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy) | At the inclusion visit on Day 0
  The investigators will record details of all patients' food allergies.
Lifestyle in Profile AMB patients (treated with non-steroidal anti-inflammatory drugs then methotrexate then biotherapy) | At the inclusion visit on Day 0
  The investigators will record details of the patient's lifestyle:
  * Brothers and sisters (number and date of birth of each one)
  * Communities (date of entry)
  * Contact with animals

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Nîmes University Hospital, Nîmes, Gard
  - Montpellier University Hospital, Arnaud de Villeneuve Hospital, Montpellier, Hérault
  - APHM, Hopital Nord, Marseille
  - Hopital des enfants, CHU de Toulouse, Toulouse